CLINICAL TRIAL: NCT00019188
Title: Phase I/II Pilot Study of Interleukin-12 in Patients With AIDS-Associated Kaposi's Sarcoma
Brief Title: Interleukin-12 in Treating Patients With AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064977; NCI-96-C-0113F; NCI-T96-0029N; NCI-MB-386; NCT00001508 (obsolete NCT alias)
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Epidemic Kaposi's Sarcoma; Recurrent Kaposi's Sarcoma
Keywords: AIDS-related malignancies; Kaposi's sarcoma; adult solid tumor; body system/site cancer; cancer; epidemic Kaposi's sarcoma; recurrent Kaposi's sarcoma; skin tumor; solid tumor; stage, Kaposi's sarcoma
MeSH Terms: conditions — AIDS-related Kaposi sarcoma; Sarcoma, Kaposi; Neoplasms; Skin Neoplasms | interventions — Interleukin-12

INTERVENTIONS:
Drug: interleukin-12

SUMMARY:
RATIONALE: Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill their tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of interleukin-12 in treating patients with AIDS -related Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of interleukin-12 (IL-12) in patients with AIDS-associated Kaposi's sarcoma.

II. Determine the antitumor activity of IL-12 in these patients. III. Determine the effect of IL-12 on angiogenic factors, including basic fibroblast growth factor, vascular endothelial growth factor, and interferon-inducible protein 10 in these patients.

IV. Determine the immunologic and virologic effects of IL-12 in these patients.

PROTOCOL OUTLINE: This is a dose escalation study. Patients receive interleukin-12 (IL-12) subcutaneously twice a week (at least 3 days apart) for 6 months. Patients with stable or better disease continue IL-12 treatment in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of IL-12 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Ten additional patients are treated at the MTD.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL:

Up to 55 patients will be entered over approximately 4.0 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically proven Kaposi's sarcoma (KS) At least 5 lesions evaluable by noninvasive methods No acutely life threatening lesions that may be responsive to other therapy Actively bleeding or critically located lesions may be excluded at the discretion of the Study Chair or Principal Investigator Asymptomatic pulmonary disease not requiring immediate cytotoxic therapy allowed HIV-associated disease Anti-HIV serum antibodies measured by ELISA and Western blot Stable dose of two or more of the following antiretroviral agents required for 4 weeks prior to study: Lamivudine Didanosine Zidovudine Saquinavir Stavudine Ritonavir Zalcitabine Indinavir Nonnucleoside reverse transcriptase inhibitor Other protease inhibitor Antiretroviral therapy unchanged during study unless medically warranted Patients may switch between antiretroviral agents provided they continue to receive a combination of 2 or more agents --Prior/Concurrent Therapy-- Biologic therapy: At least 6 months since prior interleukin-12 (IL-12) At least 3 weeks since prior interferon therapy At least 2 weeks since prior cytokines or bone marrow stimulating factors (except epoetin alfa) No concurrent cytokines except epoetin alfa or filgrastim (G-CSF) Chemotherapy: At least 3 weeks since prior chemotherapy (at least 6 weeks since prior nitrosoureas or mitomycin) At least 6 months since prior suramin Endocrine therapy: Replacement glucocorticoids allowed At least 2 months since prior systemic glucocorticoids at doses sufficient to affect immune response (e.g., more than 20 mg of prednisone or equivalent for more than 1 week) Radiotherapy: At least 3 weeks since prior radiotherapy Surgery: Not specified Other: See Disease Characteristics At least 3 weeks since prior anti-KS therapy At least 3 weeks since prior local therapy (e.g., intralesional injections) --Patient Characteristics-- Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Greater than 3 months Hematopoietic: Absolute neutrophil count at least 750/mm3 Platelet count at least 75,000/mm3 Hemoglobin at least 9.0 g/dL (no transfusion within 1 month prior to entry) Hepatic: Bilirubin no greater than 3.7 mg/dL with direct fraction no greater than 0.2 mg/dL and indirect fraction no greater than 3.5 mg/dL AST no greater than 2.5 times upper limit of normal No history of cirrhosis PT/PTT no greater than 120% of control Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 60 mL/min Other: No hypersensitivity to IL-12 or other compounds that crossreact with IL-12 No clinically significant autoimmune disease (e.g., systemic lupus erythematosus) or rheumatologic disease No active, gross gastrointestinal bleeding or uncontrolled peptic ulcer disease No inflammatory bowel disease No severe or life threatening infection with bacterial, viral, fungal, protozoal, or parasitic pathogens within 2 weeks of entry No fever of 39 degrees Celsius or higher within 10 days prior to entry unless underlying infection ruled out No second malignancy within 1 year except: Completely resected basal cell carcinoma Carcinoma in situ of the cervix No generalized debilitation or mental incapacitation that would preclude informed consent No abnormality that would score as a grade 3 toxicity other than lymphopenia or direct manifestations of KS Willing to refrain from unprotected sexual contact and other activities that could result in reinfection with HIV Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 2 months after study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 1997-01; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Medicine Branch, Bethesda, Maryland, United States